CLINICAL TRIAL: NCT02640079
Title: A Behavioral Intervention for Pain Catastrophizing in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Laura Payne, Adjunct Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001761
Record Dates: First submitted 2015-12-17; First posted 2015-12-28 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Pain Catastrophizing; Primary Dysmenorrhea
Keywords: Cognitive behavioral therapy; Laboratory pain responsivity
MeSH Terms: interventions — Cognitive Behavioral Therapy

ARMS (1):
- Cognitive behavioral therapy (Experimental): Cognitive behavioral therapy aimed at reducing pain catastrophizing.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy

SUMMARY:
The purpose of this study is to test the feasibility and efficacy of a brief group therapy treatment program focused on reducing pain catastrophizing in adolescents and young adults (ages 16-25) with menstrual pain.

ELIGIBILITY:
Inclusion Criteria:

* Female ages 16-25 years
* Self-reported menstrual cycle averaging 24-32 days
* Menstrual pain rating of ≥4 on the Numeric Rating Scale for at least the previous three menstrual cycles prior to participation
* Written informed consent or assent (if a minor, parent must also provide written parental permission)
* Able to read and understand English

Exclusion Criteria:

* Use of oral contraceptives or any exogenous hormones in the previous 3 months
* Presence of persistent pelvic pain throughout the menstrual cycle
* Acute illness or injury that may impact lab performance or that affects sensitivity of the extremities
* Diagnosis of an underlying medical cause for dysmenorrhea symptoms
* No or minimal menstrual pain (NRS rating of ≤ 3) during any of the 3 previous cycles prior to study participation
* Daily use of opioids; participants using other analgesics will be included, but will be asked not to take these analgesics on the days of the lab sessions
* Developmental delay, autism, or significant anatomic impairment that may preclude understanding of study procedures

Ages: 16 Years to 25 Years | Sex: Female
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Feasibility (as determined by attrition rate) | After each cohort completes their 5 group CBT sessions; 1 week after the 5th and final CBT session in each cohort
Acceptability - participants' views of the intervention's 1) appeal; 2) helpfulness; and 3) ease of participation | Assessed via qualitative interviews which will occur during each participant's post-intervention lab assessment (i.e., during the first two days of the first menstrual period after intervention completion)
Change in pain catastrophizing | Assessed via questionnaire completed at six time points: pre-intervention lab session, immediately following the completion of the 5th group CBT session, post-intervention lab session, and once a month for three months after intervention completion
Change in menstrual pain level assessed via 11-point numeric rating scale (NRS) | Assessed via questionnaire completed at six time points: pre-intervention lab session, immediately following the completion of the 5th group CBT session, post-intervention lab session, and once a month for three months after intervention completion
Change in medication use (dosage and frequency of pain medication use) | Assessed via questionnaire completed at six time points: pre-intervention lab session, immediately following the completion of the 5th group CBT session, post-intervention lab session, and once a month for three months after intervention completion

SECONDARY OUTCOMES:
Change in menstrual symptoms as assessed by the Menstrual Symptom Questionnaire (MSQ) | Assessed via questionnaire completed at six time points: pre-intervention lab session, immediately following the completion of the 5th group CBT session, post-intervention lab session, and once a month for three months after intervention completion
Change in anxiety as assessed by the Brief Symptom Inventory 18 (BSI-18) | Assessed via questionnaire completed at six time points: pre-intervention lab session, immediately following the completion of the 5th group CBT session, post-intervention lab session, and once a month for three months after intervention completion
Change in depression as assessed by the Brief Symptom Inventory 18 (BSI-18) | Assessed via questionnaire completed at six time points: pre-intervention lab session, immediately following the completion of the 5th group CBT session, post-intervention lab session, and once a month for three months after intervention completion
Change in somatization as assessed by the Brief Symptom Inventory 18 (BSI-18) | Assessed via questionnaire completed at six time points: pre-intervention lab session, immediately following the completion of the 5th group CBT session, post-intervention lab session, and once a month for three months after intervention completion
Change in temporal summation (TS) | Assessed at pre- and post-intervention lab sessions, each of which will occur during the first 2 days of menstruation
Change in conditioned pain modulation (CPM): pain ratings in response to a heat stimulus prior to and after administration of a conditioning pain stimulus (cold water) | Assessed at pre- and post-intervention lab sessions, each of which will occur during the first 2 days of menstruation

OTHER OUTCOMES:
Galvanic Skin Response (GSR) | Assessed at pre- and post-intervention lab sessions, each of which will occur during the first 2 days of menstruation; GSR assessed at rest (5 min), during four pain induction tasks (3-5 min each), and again at rest (5 min)
Heart Rate Variability (HRV) | Assessed at pre- and post-intervention lab sessions, each of which will occur during the first 2 days of menstruation; HRV assessed at rest (5 min), during four pain induction tasks (3-5 min each), and again at rest (5 min)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Payne, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States